CLINICAL TRIAL: NCT04118738
Title: The International Cohort Study of Children Born to Women Infected With Zika Virus During Pregnancy
Brief Title: International Cohort Study of Children Born to Women Infected With Zika Virus During Pregnancy
Status: Completed | Type: Observational
Sponsor: Westat (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Oswaldo Cruz Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ZIP 2.0
Record Dates: First submitted 2019-07-01; First posted 2019-10-08 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Zika; Neurodevelopmental Abnormality; Hearing Loss; Growth Delay; Eye Abnormalities
Keywords: ZIKA
MeSH Terms: conditions — Zika Virus Infection; Hearing Loss; Eye Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ZIKV-Exposed: Children born to women with documented confirmed or presumptive in-utero ZIKV exposure during pregnancy through delivery or the children's laboratory documentation of confirmed or presumptive in-utero ZIKV exposure within five days of birth.
- ZIKV-Unexposed: Children born to women without documented confirmed or presumptive in-utero ZIKV exposure during pregnancy through delivery and the children have no laboratory documentation of confirmed or presumptive in-utero ZIKV exposure at any time prior to ZIP 2.0 enrollment, if testing was performed prior to enrollment.

SUMMARY:
The International Cohort Study of Children Born to Women Infected with Zika Virus (ZIKV) During Pregnancy study is a prospective, observational, international cohort study of children previously enrolled in the ZIP study or other ZIP 2.0 Protocol Team approved ZIKV-cohort study that will continue the longitudinal follow-up of children born with documented confirmed or presumptive in-utero ZIKV exposure ("ZIKV-exposed" cohort) and children born without documented confirmed or presumptive in-utero ZIKV exposure, matched by site and birth sex ("ZIKV-unexposed" cohort).

Follow-up evaluations and assessments will allow for the determination and comparison of long-term neurodevelopmental outcomes among in utero ZIKV-exposed and ZIKV-unexposed children. Each participant will be followed for about 2 years, beginning at approximately 18 months through 42 months of age.

DETAILED DESCRIPTION:
The International Prospective Observational Cohort Study of Zika in Infants and Pregnancy (ZIP) study has leveraged 10 international sites to follow mother-infant dyads prospectively in pregnancy and postpartum to determine the incidence and outcomes of Zika Virus (ZIKV) infection. The ZIP study has collected demographic, physical, environmental, laboratory, and delivery outcome data in relation to mother-infant pairs with and without ZIKV infection. Infants born to women enrolled in the ZIP study are followed for 1 year and undergo regular physical and neurological assessments to identify clinical or developmental outcomes.

The International Cohort Study of Children Born to Women Infected with Zika Virus During Pregnancy (ZIP 2.0) study will enroll children who themselves or whose biological mothers were previously enrolled in the ZIP study and other ZIP 2.0 Protocol Team-approved studies. Assessments include growth, neurodevelopmental, audiologic, ophthalmologic, and other clinical outcomes. Evaluations will occur about every 6 months over about a 2-year period beginning at approximately 18 months of age. Follow-up evaluations and assessments will allow for the determination and comparison of long-term neurodevelopmental outcomes among in utero ZIKV-exposed and ZIKV-unexposed children.

After parent(s)/legal guardian(s) permission is obtained for the child's participation in ZIP 2.0, several means to contact them will be requested. Parents will be asked whether or not messages can be left for each of the phone numbers provided and if messages can contain information regarding the nature of the study.

We expect to compare approximately 200 children with documented confirmed or presumptive in-utero ZIKV exposure and 200 controls matched by site and birth sex without documented confirmed or presumptive in-utero ZIKV exposure at age approximately 18 months, and at age 42 months.

The primary objective is to determine the long-term neurodevelopmental outcomes among children born with documented confirmed or presumptive in-utero ZIKV exposure. The secondary objectives are to compare the long-term effects (e.g., on growth, vision, hearing and neurodevelopment) of in-utero ZIKV-exposure compared to unexposed children.

ELIGIBILITY:
Inclusion Criteria:

ZIKV- Exposed Inclusion Criteria:

* Parent(s)/legal guardian(s) provided written permission for his or her child to participate.
* Participant and/or participant's biological mother previously enrolled in the ZIP study or other ZIKV cohort study approved by the sponsors.
* Participant's biological mother has laboratory documentation of positive ZIKV RNA test results during pregnancy through delivery delivery or the participant has laboratory documentation of ZIKV RNA or serology positive/presumptive positive/equivocal ZIKV test within 5 days of birth according to the ZIKV-exposed definitions included in the ZIP 2.0 inclusion criteria.
* Minimum 74 weeks of age (approximately 17months) of age at enrollment

ZIKV-Unexposed Inclusion Criteria:

* Parent(s)/legal guardian(s) provided written permission for his or her child to participate.
* Previously enrolled in the ZIP study and identified as matching the same birth sex and followed at the same study site as an enrolled ZIKV-exposed participant.
* Laboratory documentation that the participant's biological mother has negative ZIKV RNA test results and no positive ZIKV RNA test results at any time during her pregnancy through delivery.
* Participant did not test ZIKV RNA and/or serology positive presumptive positive or equivocal at any time prior to ZIP 2.0 enrollment, if testing was performed prior to enrollment.
* Minimum 74 weeks of age (approximately 17months) of age at enrollment

Exclusion Criteria: Both Exposed and Unexposed Cohorts

• Enrolled in other clinical research (including other ZIKV research) requiring blood collection, which in combination with ZIP 2.0 evaluations, would exceed the lesser of 50 mL or 3 mL per kg in an 8-week period and/or blood collection would be required more frequently than two times per week.

Ages: 18 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Approximately 200 children with confirmed or presumptive in-utero exposure to Zika virus and approximately 200 children matched by site and birth sex without confirmed or presumptive in-utero exposed to Zika virus.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental outcome at age18 months | At enrollment
  Neurodevelopment will be measured at age 18 months (entry visit) with the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III). The scores indicates how well the child performed compared to a group of children within the same age range.
Neurodevelopmental outcome at age 24 months | Six months after enrollment
  Neurodevelopment will be measured at age 24 months with the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III).
Neurodevelopmental outcome at age 30 months | Twelve months after enrollment
  Neurodevelopment will be measured at age 30 months with the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III).
Neurodevelopmental outcome at age 36 months | Eighteen months after enrollment.
  Neurodevelopment will be measured at age 36 months with the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III).
Neurodevelopmental outcome at age 42 months | Twenty four months after enrollment
  Neurodevelopment will be measured at age 42 months with the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III).

SECONDARY OUTCOMES:
Anthropometric Measurements: Height | At enrollment
  Height in centimeters will be measured at age 18 months (entry visit).
Anthropometric Measurements: Height | Six months after enrollment
  Height in centimeters will be measured at age 24 months
Anthropometric Measurements: Height | Twelve months after enrollment
  Height in centimeters will be measured at age 30 months
Anthropometric Measurements: Height | Eighteen months after enrollment
  Height in centimeters will be measured at age 36 months
Anthropometric Measurements: Height | Twenty-four months after enrollment
  Height in centimeters will be measured at age 42 months
Anthropometric Measurements: Weight | At enrollment
  Weight in kilograms will be measured at age 18 months (entry visit).
Anthropometric Measurements: Weight | Six months after enrollment
  Weight in kilograms will be measured at age 24 months (entry visit).
Anthropometric Measurements: Weight | Twelve months after enrollment
  Weight in kilograms will be measured at age 30 months (entry visit).
Anthropometric Measurements: Weight | Eighteen months after enrollment
  Weight in kilograms will be measured at age 36 months (entry visit).
Anthropometric Measurements: Weight | Twenty-four months after enrollment
  Weight in kilograms will be measured at age 42 months (entry visit).
Anthropometric Measurements: Head circumference | At enrollment
  Head circumference in centimeters will be measured at age 18 months (entry visit).
Anthropometric Measurements: Head circumference | Six months after enrollment
  Head circumference in centimeters will be measured at age 24 months.
Anthropometric Measurements: Head circumference | Twelve months after enrollment
  Head circumference in centimeters will be measured at age 30 months.
Anthropometric Measurements: Head circumference | Eighteen months after enrollment
  Head circumference in centimeters will be measured at age 36 months.
Anthropometric Measurements: Head circumference | Twenty-four months after enrollment
  Head circumference in centimeters will be measured at age 42 months.
Anthropometric Measurements: Mid upper arm circumference | Six months after enrollment
  Mid upper arm circumference in centimeters will be measured at age 24 months
Anthropometric Measurements: Mid upper arm circumference | At enrollment
  Mid upper arm circumference in centimeters will be measured at age 18 months
Anthropometric Measurements: Mid upper arm circumference | Twelve months after enrollment
  Mid upper arm circumference in centimeters will be measured at age 30 months
Anthropometric Measurements: Mid upper arm circumference | Eighteen months after enrollment
  Mid upper arm circumference in centimeters will be measured at age 36 months
Anthropometric Measurements: Mid upper arm circumference | Twenty-four months after enrollment
  Mid upper arm circumference in centimeters will be measured at age 42 months
Hearing assessment: A-verage (in dB HL) of the value of Air-conduction test obtained for all frequencies measured (500Hz, 1000 Hz, 2000Hz and 4000Hz).Audiometry (VRA) | At enrollment (visit 1) only if the participant missed the evaluation(s) at the 12-month ZIP study visit or is 95 or greater weeks of age at the Entry visit; then, six months after enrollment (visit 2), and 18 months after enrollment (visit 4).
Hearing assessment: Average (in dB HL) of Bone-conduction test obtained for all frequencies measured (500Hz, 1000 Hz, 2000Hz and 4000Hz). | At enrollment (visit 1) only if the participant missed the evaluation(s) at the 12-month ZIP study visit or is 95 or greater weeks of age at the Entry visit; then, six months after enrollment (visit 2), and 18 months after enrollment (visit 4).
Hearing assessment: Proportion of children in different categories of the degree of hearing loss | At enrollment (visit 1) only if the participant missed the evaluation(s) at the 12-month ZIP study visit or is 95 or greater weeks of age at the Entry visit; then, six months after enrollment (visit 2), and 18 months after enrollment (visit 4).]
  Proportion of children in different categories of the degree of hearing loss (Normal hearing; Mild hearing loss; Moderate hearing loss; Severe hearing loss; and Profound hearing loss). The degree of hearing loss will be determined by grouping the average of the value of Air-conduction test obtained for all frequencies measured (500Hz, 1000 Hz, 2000Hz and 4000Hz).
Hearing assessment: Proportion of children in different categories of the type of hearing loss | At enrollment (visit 1) only if the participant missed the evaluation(s) at the 12-month ZIP study visit or is 95 or greater weeks of age at the Entry visit; then, six months after enrollment (visit 2), and 18 months after enrollment (visit 4).]
  Proportion of children in different categories of the type of hearing loss (Sensorineural hearing loss; Conductive hearing loss; and Mixed hearing loss). The type of hearing loss will be established by comparing the mean of air-conduction levels.
Hearing assessment: Proportion of children with abnormal results in the Otoacustic Emissions test. | Time Frame: At enrollment only if the participant missed the evaluation(s) at the 12-month ZIP study visit or is 95 or greater weeks of age at the Entry visit; then, six months after enrollment, and 18 months after enrollment.
Comprehensive ophthalmologic evaluation. | At enrollment (visit 1) only if the participant missed the evaluation(s) at the 12-month ZIP study visit or is 95 or greater weeks of age at the Entry visit; then, six months after enrollment (visit 2), and 18 months after enrollment (visit 4).
  General examination of eye structure and assessment of visual function. Composite measure of Visual function based on visual behaviors (with minimum and maximum possible values of -6 and +6, respectively).
Comprehensive ophthalmologic evaluation | At enrollment (visit 1) only if the participant missed the evaluation(s) at the 12-month ZIP study visit or is 95 or greater weeks of age at the Entry visit; then, six months after enrollment (visit 2), and 18 months after enrollment (visit 4)
  Composite measure of Retina evaluation (with minimum and maximum possible values of -14 and +14, respectively).
Comprehensive ophthalmologic evaluation | At enrollment (visit 1) only if the participant missed the evaluation(s) at the 12-month ZIP study visit or is 95 or greater weeks of age at the Entry visit; then, six months after enrollment (visit 2), and 18 months after enrollment (visit 4).]
  Composite measure of Optic Nerve evaluation (with minimum and maximum possible values of -12 and +12, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Deolinda MF Scalabrin, MD, PhD, Study Chair — Research Center- FIOCRUZ Brazil; Marisa M. Mussi-Pinhata, MD, MD, Study Chair — Ribeirão Preto Medical School- University of Sao Paulo; Maria Elisabeth L Moreira, MD, Study Chair — Instituto Fernandes Figueira - FIOCRUZ
Locations (5):
- Brazil (2):
  - Departamento de Medicina Tropical da Universidade Federal de Pernambuco- UFPE, Recife, Pernambuco
  - Instituto Fernandes Figueira - FIOCRUZ, Rio de Janeiro
- Centro Médico Imbanaco (CMI), Cali, Colombia
- Asociación Civil Selva Amazónica, Iquitos, Loreto, Peru
- Puerto Rico Medical Center- Maternal Infant Studies Center (CEMI), San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided